CLINICAL TRIAL: NCT03763344
Title: An Examination of Visual Perceptual Training in Older Adults With Subjective Memory Complaints
Brief Title: An Examination of Visual Perceptual Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Victoria (Other)
Responsible Party: Principal Investigator, Brian Christie, Professor, CIHR Delegate and Health Research Advisory Committee Chair Division of Medical Sciences,, University of Victoria
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 19-123
Record Dates: First submitted 2018-10-22; First posted 2018-12-04 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Age-Related Memory Disorders
Keywords: memory; visual spatial training; multiple object tracking; Elderly
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort C (Experimental): Older adults over the age of 60 years old with subjective memory complaints that underwent:
  * the first cognitive assessment (Baseline),
  * intervention is fourteen sessions of Perceptual Cognitive Training (PCT) for seven weeks,
  * a post-treatment cognitive assessment (Week 7), and
  * a follow up cognitive assessment (Week 11)
  Interventions: Behavioral: Perceptual Cognitive Training (PCT)
- Cohort D (No Intervention): Older adults over the age of 60 years old with subjective memory complaints that underwent:
  * the first cognitive assessment (baseline),
  * seven weeks of no intervention,
  * a post-treatment cognitive assessment (week 7), and
  * a follow up cognitive assessment (week 11)

INTERVENTIONS:
Behavioral: Perceptual Cognitive Training (PCT) — Perceptual Cognitive Training (PCT) will be performed by having individuals work with a visual perceptual training software program called NeuroTracker. This device uses Multiple Object Tracking at increasing difficulties to develop high-level brain functions critical to recovery & cognitive health. By increasing in difficulty with each correct response and decreasing in difficulty when mistakes are made, brain function is constantly challenged. Each session (6 mins) delivers a series of mini-tests where the patient needs to remember key targets, then track them moving among distractors for several seconds and then identify them. Simple to do, but always challenging, NeuroTracker adaptively optimizes difficulty to each patient's level, maximizing cognitive stimulation every step of the way.
  Arms: Cohort C

SUMMARY:
Perceptual-cognitive training (PCT) is a computerized software game has been shown to improve sport performance in young elite athletes and even to aid in recovery speeds post-concussion. PCT may represent a unique type of training that could ultimately enhance cognitive performance or quality of life in all populations. What is not clear is whether PCT is beneficial to older adults with subjective memory complaints (SMCs). SMCs in older adults are an early risk indicator for Alzheimer's disease, making older adults with SMCs a target population for proactive interventions. The aim of this study was to determine if PCT can serve as a proactive intervention and enhance cognitive abilities in older adults with SMCs. The results of this research protocol introduce a new way of prevention from cognitive decline in healthy older adults and may introduce a new training programs for age-related memory disorder.

DETAILED DESCRIPTION:
This study was approved by the University of Victoria Human Research Ethics Board (Protocol Number 17-167) and all participants provided their informed written consent prior to participating in this study. In order to reduce the placebo effect, the participants were randomly divided into the experimental and control groups. Participants from both the experimental and control groups received a total of three neuropsychological assessments over a three month period (i.e. baseline, 7 weeks, 11 weeks). Considering that an essential methodological component of the training studies is the use of standardized neuropsychological tests, validated and reliable measures such as STROOP TEST, DIGIT SPAN TEST, TRAIL MAKING TEST, VERBAL FLUENCY TESTS, CALIFORNIA VERBAL LEARNING TEST Second Edition (i.e., standard and alternate forms), were used at different time points. Each assessment was 50-60 minutes in duration and was administered by an expert neuropsychology resident. The first assessment was administered at baseline . Then, the experimental group underwent seven weeks of perceptual cognitive training, while the control group completed seven weeks without formal training. The treatment for the PCT group consisted of 14 sessions of training each lasting 25-30 min, twice per week for seven weeks. After the seven-week time period, a second neuropsychological assessment was performed on both groups. After eleven weeks, a follow-up assessment was conducted to verify whether the benefits of cognitive training endure over time.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 and over;
* Have subjective cognitive complaints;
* The results of the screening test Mini Mental State Examination (MMSE) should be ≥ 24 (this test is used only at baseline visit to verify if the participant might be included in the sample or not).

Exclusion Criteria:

* Presence of medical diagnosis of a Major Neurocognitive Disorder (e.g. Alzheimer's disease, front temporal lobe dementia, Lewy Body dementia, vascular dementia),
* Presence of sensory deficits (e.g. colour blindness, monocular/binocular blindness, macular degeneration),
* Presence of psychiatric disorders (i.e. depression, anxiety),
* The participants with scores under 24 at MMSE screening test will be excluded and sent to the family doctor (i.e. to minimize the risk of including people with pre-clinical dementia).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-15 (Actual)

PRIMARY OUTCOMES:
Change in memory performance in older adults with SMCs | First neuropsychological assessment (Baseline). After seven week period both groups underwent the second neuropsychological assessment (Week 7). After eleven weeks a follow-up assessment was conducted (Week 11).
  Assessed by CALIFORNIA VERBAL LEARNING TEST

SECONDARY OUTCOMES:
Change in processing speed in older adults with SMCs | First neuropsychological assessment (Baseline). After seven week period both groups underwent the second neuropsychological assessment (Week 7). After eleven weeks a follow-up assessment was conducted (Week 11).
  Assessed by Delis-Kaplan Executive Function System™ (D-KEFS™).
Change in cognitive flexibility in older adults with SMCs | First neuropsychological assessment (Baseline). After seven week period both groups underwent the second neuropsychological assessment (Week 7). After eleven weeks a follow-up assessment was conducted (Week 11).
  Assessed by Delis-Kaplan Executive Function System™ (D-KEFS™)
Change in cognitive flexibility in older adults with SMCs | First neuropsychological assessment (Baseline). After seven week period both groups underwent the second neuropsychological assessment (Week 7). After eleven weeks a follow-up assessment was conducted (Week 11).
  Assessed by Stroop Test
Change in working memory in in older adults with SMCs | First neuropsychological assessment (Baseline). After seven week period both groups underwent the second neuropsychological assessment (Week 7). After eleven weeks a follow-up assessment was conducted (Week 11).
  Assessed by Digit Span Test

CONTACTS AND LOCATIONS:
Overall Officials: Brian R. Christie, Ph.D, Principal Investigator — University of Victoria
Locations (1):
- University of Victoria, Victoria, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berry AS, Zanto TP, Clapp WC, Hardy JL, Delahunt PB, Mahncke HW, Gazzaley A. The influence of perceptual training on working memory in older adults. PLoS One. 2010 Jul 14;5(7):e11537. doi: 10.1371/journal.pone.0011537. PMID 20644719
- [Background] Anguera JA, Boccanfuso J, Rintoul JL, Al-Hashimi O, Faraji F, Janowich J, Kong E, Larraburo Y, Rolle C, Johnston E, Gazzaley A. Video game training enhances cognitive control in older adults. Nature. 2013 Sep 5;501(7465):97-101. doi: 10.1038/nature12486. PMID 24005416
- [Background] Cavanagh P, Alvarez GA. Tracking multiple targets with multifocal attention. Trends Cogn Sci. 2005 Jul;9(7):349-54. doi: 10.1016/j.tics.2005.05.009. PMID 15953754
- [Background] Parsons B, Magill T, Boucher A, Zhang M, Zogbo K, Berube S, Scheffer O, Beauregard M, Faubert J. Enhancing Cognitive Function Using Perceptual-Cognitive Training. Clin EEG Neurosci. 2016 Jan;47(1):37-47. doi: 10.1177/1550059414563746. Epub 2014 Dec 30. PMID 25550444
- [Background] Tullo D, Guy J, Faubert J, Bertone A. Training with a three-dimensional multiple object-tracking (3D-MOT) paradigm improves attention in students with a neurodevelopmental condition: a randomized controlled trial. Dev Sci. 2018 Nov;21(6):e12670. doi: 10.1111/desc.12670. Epub 2018 Apr 30. PMID 29707864
- [Background] Faubert J. Visual perception and aging. Can J Exp Psychol. 2002 Sep;56(3):164-76. doi: 10.1037/h0087394. PMID 12271747